CLINICAL TRIAL: NCT04672122
Title: The Effects of Cathodal tDCS on Muscle Strength in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: MU-CIRB2020/314.0210
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation (tDCS) will be applied for 20 mins. Cathode on the primary motor area (M1) and Anode on the supraorbital area of contralateral side. Current intensity will be at 2 mA (sham mode). The scope of intervention is to investigate effect of sham tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal-tDCS 1 mA (Experimental): Cathodal transcranial direct current stimulation (tDCS) will be applied for 20 mins. Cathode on the primary motor area (M1) and Anode on the supraorbital area of contralateral side. Current intensity is fixed at 1 mA and current will flow continuously. The scope of intervention is to investigate effect of cathodal tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal-tDCS 1.5 mA (Experimental): Cathodal transcranial direct current stimulation (tDCS) will be applied for 20 mins. Cathode on the primary motor area (M1) and Anode on the supraorbital area of contralateral side. Current intensity is fixed at 1.5 mA and current will flow continuously. The scope of intervention is to investigate effect of cathodal tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal-tDCS 2 mA (Experimental): Cathodal transcranial direct current stimulation (tDCS) will be applied for 20 mins. Cathode on the primary motor area (M1) and Anode on the supraorbital area of contralateral side. Current intensity is fixed at 2 mA and current will flow continuously. The scope of intervention is to investigate effect of cathodal tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Cathodal tDCS will be applied for 20 mins.

SUMMARY:
To investigate the effects of different intensity of cathodal tDCS on muscle strength in healthy adults.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate cortical excitability. In 2000, Nitsche and Paulus reported the polarity-dependent effect of tDCS in humans, i.e., anodal tDCS facilitates cortical excitability while cathodal tDCS decreases it. (Nitsche & Paulus, 2000). TDCS studies have been replicated by many researchers and reported similar effects of tDCS in humans when using anodal and cathodal tDCS with an intensity of 1 mA. The linear effect of tDCS also has been reported by various studies, i.e., when increase intensity, the polarity-dependent effect of tDCS also enhances. However, conflicting results of cathodal tDCS efficacy have been reported.

Cortical excitability has been used to represent the efficacy of tDCS on neuroplasticity. The linear effect of cathodal tDCS on cortical excitability have been reported by researchers when using intensities at 1, 2, and 3 mA stimulated at the primary motor cortex in healthy participants (Batsikadze et al., 2013; Jamil et al., 2017; Kuo et al., 2013; Mosayebi Samani et al., 2019; Nitsche et al., 2003). Nevertheless, some studies showed the non-linear effects of cathodal tDCS (i.e., when increases intensity, cathodal tDCS enhances the cortical excitability) when using intensities at 1.5 and 2 mA in healthy participants (Batsikadze et al., 2013; Jamil et al., 2017; Mosayebi Samani et al., 2019). Hence, cathodal tDCS efficacy on cortical excitability is still controversy.

Muscle performance is an outcome that represents clinical change induced by tDCS. Previous studies reported the tendency of cathodal tDCS efficacy in decreasing muscle performance of both upper and lower extremities in healthy participants (Cogiamanian et al., 2007; Tanaka et al., 2009). However, previous studies used a single intensity of tDCS in each study. Hence, there was no direct comparison between different intensities of cathodal tDCS on muscle performance in healthy participants.

In our study, we aim to investigate the effect of different intensities of cathodal tDCS on muscle strength in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy adults
2. Age range between 18 - 60 years old
3. Right-handed dominant identified by the Edinburg Handedness Inventory
4. No recent muscle injuries of both limbs for a past 6-months

Exclusion Criteria:

1. Consumed caffeine within 24 hours prior the experiment
2. History of neurological symptoms i.e. seizures, weakness, loss of sensation or unclear history of pass illness
3. Presence of metal implantation, intracranial shunt, cochlear implantation or cardiac pacemakers
4. Presence of opened wound or infectious wound around scalp
5. Presence of pain in evaluating muscle groups
6. History of surgery in evaluating limbs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline muscle strength after tDCS | Baseline (Pretest) and 40 minutes ( posttest)
  Muscle strength will be measured in Newton by using a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vimolratana O, Lackmy-Vallee A, Aneksan B, Hiengkaew V, Klomjai W. Non-linear dose response effect of cathodal transcranial direct current stimulation on muscle strength in young healthy adults: a randomized controlled study. BMC Sports Sci Med Rehabil. 2023 Jan 30;15(1):10. doi: 10.1186/s13102-023-00621-7. PMID 36717894